CLINICAL TRIAL: NCT03931889
Title: Effects of Vitamin D3 Supplementation on Antioxidant Enzymes Status in Vitamin D3 Deficient Asthma COPD Overlap (ACO) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr.Maksuda Bintey Mahmud, MD course student, Department of Physiology,BSMMU,Dhaka,Bangladesh, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BSMMU/2018/6813
Record Dates: First submitted 2019-04-22; First posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D3 (Active Comparator): Cholecalciferol 80,000 IU (2 capsules of 40,000 IU) per oral per week for consecutive 26 weeks.
  Interventions: Dietary Supplement: Vitamin D3
- Vitamin D3 placebo (Placebo Comparator): Placebo (2 capsules) per oral per week for consecutive 26 weeks.
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Cap. Cholecalciferol 40,000 IU

SUMMARY:
Asthma-COPD overlap (ACO) is a new entity in the world of respiratory ailments. The respiratory tract of these patients are continuously exposed to oxidants (due to cigarette smoking) causing oxidative stress. Antioxidant enzymes such as, superoxide dismutase (SOD) and catalase (CAT) neutralize these oxidants or free radicals and transform them into safer. Vitamin D is a natural antioxidant which has few evidence of increasing antioxidant enzyme level in COPD and asthma, but not in ACO patients. To evaluate the effects of vitamin D3 supplementation on antioxidant enzymes level in vitamin D3 deficient patients with stable ACO. The randomized controlled trial was conducted in Department of Physiology Bangabandhu Sheikh Mujib Medical University (BSMMU), Shahbag, Dhaka from March 2018 to February 2019. For this study, a total number of 40 vitamin D3 deficient (serum 25 hydroxycholecalceferol <30 ng/ml) male, stable (diagnosed patient, who was not experienced any acute exacerbation, hospitalization, urgent care visits or changes in routine medication within 4 weeks prior to study) patients with ACO of age ≥40 years was selected from the Out Patient Department (OPD) of the National Institute of Diseases of Chest and Hospital (NIDCH) and randomly grouped as A (control) and B (study). Then serum Superoxide dismutase and Catalase level of all the patients was assessed. Along with the standard pharmacological treatment of ACO (according to GOLD criteria), oral vitamin D3 (80,000 IU per week) will be supplied to the patients of the 'Study group' and placebo for 'Control group' for consecutive 26 weeks. At 26th week of follow up, all the study variables were examined. With this, all patients of both the groups were advised to continue ad lib (according to their own choice) diet. The results was expressed as mean±SD and the data was statistically analyzed by SPSS Version 16, using Independent sample 't' test (between two groups) and paired student's 't' test (between paired groups before and after intervention). In the interpretation of results, <0.05 level of probability (p) was accepted as significant.

ELIGIBILITY:
Inclusion Criteria:

* Smoker
* Stable ACO patients
* Vitamin D3 deficieny
* Duration of ACO: 1-4 years

Exclusion Criteria:

* With acute exacerbation of any pulmonary diseases, as- respiratory tract infection, bronchiectasis,pleural effusion,tuberculosis, interstitial lung disease, pneumonectomy or pulmonary lobectomy.
* Any cardiac disease.
* Chronic liver disease
* Malignancy
* Use of drugs within 1 month prior to study, as- calcium supplement, Phenytoin, Carbamazepine, Clotrimazole, Rifampicin, Nifedipine, Spironolactone, Ritononavir, Saquinavir, Cyproterone acetate, glucocorticoids, bisphosphonate
* With biochemical evidence of - uncontrolled diabetes mellitus, renal insufficiency

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Plasma Superoxide dismutase (SOD) level | 26th week of vitamin D3 supplementation
  Plasma Superoxide dismutase (SOD) after 26 weeks of vitamin D3 supplementation
Plasma Catalase (CAT) level | 26th week of vitamin D3 supplementation
  Plasma Catalase (CAT) after 26 weeks of vitamin D3 supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Taskina Ali, MBBS,M.Phil, Study Director — BSMMU, Shahbagh, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University (BSMMU), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No